CLINICAL TRIAL: NCT05731297
Title: Perineal, Psychological and Well-beeing Consequences of Conflict-related Sexual Violence Among Women Living in Democratic Republic of Congo
Brief Title: Consequences of Sexual Violence Among Women Living in Democratic Republic of Congo
Acronym: SV-RDC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bertuit Jeanne (Other)
Collaborators: University of Kinshasa (Other)
Responsible Party: Sponsor-Investigator, Bertuit Jeanne, Principal Investigator, University of Applied Sciences of Western Switzerland
Organization: University of Applied Sciences of Western Switzerland (Other)
Other Study IDs: 2021-01
Record Dates: First submitted 2023-01-20; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Sexual Violence; Woman Abuse; Perineal Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women victims of CRSV: * Inclusion criteria: Women victims of CRSV living in the places of enrolment in RDC, aged over 18 years and giving their consent to participate to this study.
  * Exclusion criteria: Pregnant women and women under 18 years old.
- women without a history of CRSV: * Inclusion criteria: women without a history of CRSV living in the places of enrolment in RDC, aged over 18 years and giving their consent to participate to this study.
  * Exclusion criteria: Pregnant women and women under 18 years old.

SUMMARY:
In conflict situations, sexual violence (SV) used can take various forms, including rape and female genital mutilation (FGM). SV is used as a strategic weapon to shake, terrorize, and displace communities and thus take control of a particular population or territory. For two decades, the Great Lakes region of Central Africa, which includes the eastern part of the Democratic Republic of the Congo (DRC), has experienced a high degree of instability due to various armed conflicts. The attacks on civilians are illustrated by SV. In 2011, studies in DRC estimated that 1 150 women are raped every day and that 30% of women have experienced conflict-related sexual violence (CRSV) over the past 16 years. In addition to physical suffering, survivors of CRSV must live with psychological consequences. Traumatic fistula, one of the most extreme consequences of SV, is well described in the literature, as its surgical management. In contrast, the literature and the government illustrate a lack of accurate data on the physical consequences such as pelvic dysfunction and psychologic disorders following these attacks. To be able to put in place adequate care, it is necessary to identify the conditions and needs of the victims.

DETAILED DESCRIPTION:
The project to collaborate with the DRC is initiated from an ambition of the pelvic-perineal rehabilitation unit of the Department of Physical Medicine and Rehabilitation (Faculty of Medicine, University of Kinshasa) to change the situation in relation to women and to be able to offer adequate care for this population. The project is part of collaboration with two investigators: Professor Miangindula (Université de Kinshasa, UNIKIN) in DRC and Professor Bertuit (HESAV-HES-SO) in Lausanne (Switzerland). Four partners will take part in the project enabling a competent and strong team: Professor Feipel and Professor Foucart (Université Libre de Bruxelles, ULB) in Brussels (Belgium), Doctor Abdulcadir (Hôpital Universitaire de Genève, HUG) and Professor Mukwege in Bukavu (DRC). This project pursues two objectives: firstly, to assess clinical data of pelvic floor dysfunction (pelvic floor muscle function and urinary, sexual, gynaecological, and anal function) and psychological level in women victims of CRSV compared to women not victims of CRSV in the DRC. Secondly, to investigate the current care modalities and to analyse their needs (access to care, community integration, physiotherapy, etc.) and to understand the global context of care in DRC. The project will contribute to scientific capacity building by involving two PhD students in this research. A mixed method research will include a quantitative design, an observational study in a sample of women victims of CRSV (n = 371) and a control group of women not victims of CRSV (n = 371). Outcomes on urinary, sexual, gynaecological, anorectal and psychological aspects will be collected. This study includes a qualitative study with a phenomenological approach. Individual semi-structured interviews will be conducted with women victims of CRSV (n=10). Interview topics will be complemented with quantitative data and will lead to the following themes: experiences of CRSV, consequences of CRSV on body image, and modalities and needs for caring of these consequences. Two focus groups including eight medical health professionals will complete the qualitative data collection. The project will be realized over three years in the most affected provinces of the DRC: South and North Kivu. The method for cross-referencing data will be the Sequential Explanatory Method described by Creswell (2013).

ELIGIBILITY:
Inclusion Criteria:- Women victims of CRSV and women without a history of CRSV living in the places of enrolment in RDC, aged over 18 years and giving their consent to participate to this study.

-

Exclusion Criteria:- Pregnant women and women under 18 years old.

-

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women in RDC
Sampling Method: Non-Probability Sample
Enrollment: 742 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Urinary aspects | At the test time
  Urinary aspects will be assessed by one questionnaire: International Consultation on Incontinence Questionnaire Female Lower Urinary Tract SymptomsModules (ICIQ-FLUTS)
Sexual aspects | At the test time
  Sexual aspects will be assessed by one questionnaire: Female Sexual Function Index (FSFI)
Pelvic and Perineal aspect | At the test time
  Pelvic and Perineal aspect will be assessed by clinical examination made by a women assistant of the research team, physiotherapist expert on pelvic floor field • Examen of observation: presence of scars, lesions, inflammation, type of FGM as described by WHO classification and types of scars during external exam; Perineal pain, intensity and localization with Haslam and Laycock ring of continence, pelvic floor muscle tone with the Reissing tone scale which have a good interrater reliability for intra-vaginal manual assessment of pubococcygeus tone for expert examinator. Laycock's power, endurance, repetitions, fast contractions, every contraction timed (PERFECT) scale will be used for pelvic floor muscle assessment. The PERFECT scheme has demonstrated good reliability and validity as an assessment tool.
  .
Ano-rectal aspect | At the test time
  Two questionnaires will be used; one to assess anal incontinence (AI) and one for constipation
  * The St. Mark's Incontinence Score (SMIS)
  * The Knowles, Eccersley, Scott Symptom Score (KESS

SECONDARY OUTCOMES:
Psychological aspect: will assessing with be PCL-5 questionnaire | At the test time
  Psychological aspect: will assessing with be PCL-5 questionnaire The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5)
Quality of Life (QoL) | At the test time
  The Medical Outcomes Study MOS 36-Item Short Form Health Survey (SF-36)

OTHER OUTCOMES:
Sociodemographic characteristic data | At the test time
  Sociodemographic characteristic data will be collected with the following variables: age, marital status, the number of pregnancies, presence of traditional genital mutilation, presence of sexual violence and CRSV (age of aggression, type of sexual violence, the moment and number of sexual violence and aggressors), education, residence, parity, nationality and tribes.

CONTACTS AND LOCATIONS:
Locations (1):
- Betty Miangindula, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided